CLINICAL TRIAL: NCT02633384
Title: Incidence and Severity of Parenteral Nutrition Associated Cholestasis in Neonates Subjected to Major Surgery, Using Two Mixed Intravenous Lipid Emulsions
Brief Title: Reduction of Neonatal Parenteral Nutrition Associated Cholestasis Through Lipid Emulsions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: One of the intravenous lipid emulsions was retired from the market
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Principal Investigator, Luís Pereira-da-Silva, MD, PhD, Centro Hospitalar de Lisboa Central
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHLC.CI70.2014
Record Dates: First submitted 2015-11-30; First posted 2015-12-17 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Intrahepatic, Cholestasis
Keywords: Parenteral nutrition associated cholestasis; Intravenous lipid emulsions; Surgical neonates; Congenital gastrointestinal abnormalities
MeSH Terms: conditions — Cholestasis, Intrahepatic | interventions — SMOFlipid; Lipofundin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMOFlipid (Experimental): infants subjected to corrective surgery for congenital abnormalities and needing prolonged PN using a new generation intravenous lipid emulsion
  Interventions: Other: SMOFlipid
- Lipofundin (Other): infants subjected to corrective surgery for congenital abnormalities and needing prolonged PN using a current intravenous lipid emulsion
  Interventions: Other: Lipofundin

INTERVENTIONS:
Other: SMOFlipid — Exclusive total parenteral nutrition using a new generation intravenous lipid emulsion composed of 30% LCT n-6 (soybean oil), 30% MCT (coconut oil), 25% monounsaturated fatty acids (olive oil), 15% LCT n-3 (fish oil) and α-tocopherol
  Other Names: SMOFlipid® (Fresenius Kabi)
  Arms: SMOFlipid
Other: Lipofundin — Exclusive total parenteral nutrition using a current intravenous lipid emulsion composed of 50% LCT (soybean oil) and 50% MCT (coconut oil)
  Other Names: Lipofundin® (B Braun)
  Arms: Lipofundin

SUMMARY:
Parenteral nutrition associated cholestasis (PNAC) is a common complication of prolonged and exclusive parenteral nutrition (PN). Infants subjected to major surgery are often unable to receive enteral nutrition for a long period of time, during which they require exclusive PN. In preterm infants, hepatic immaturity is a predisposing factor. Intravenous lipid emulsions (ILE) used in PN may promote PNAC or protect against it depending on their composition. Medium chain triglycerides (MCT) may have a hepatic protective effect. Long chain triglycerides (LCT) of n-3 family may protect from PNAC. In several new-generation emulsions, the α-tocopherol content is higher than the gamma-tocopherol content, acting as an antioxidant, preventing lipid peroxidation.

The incidence and severity of PNAC in term and near-term infants subjected to corrective surgery for congenital abnormalities and needing prolonged PN using the ILE SMOFlipid® or Lipofundin® is compared. The investigators hypothesise that SMOFlipid® is more protective from PNAC than Lipofundin®.

Single-center, randomized, controlled and double-blinded trial on consecutive neonates admitted in the NICU, with gestational age of 34 weeks or over, undergoing corrective surgery of congenital anomaly of the digestive tract or indirectly affecting the digestive tract. Recruitment if PN with ILE was started within the first 48 hours after birth. Minimum intervention: exclusive PN for at least 1 week.

Main outcome: incidence of cholestasis (conjugated serum bilirubin >1 mg/dl [34 mmol/L]). Severity of cholestasis evaluated by the magnitude of the serum conjugated bilirubin and serum γ-glutamyltranspeptidase (GGT). Mixed effects regression models are used to take into account the correlation structure between measures in time. Crude and adjusted odds-ratios with corresponding 95% confidence intervals are calculated.

DETAILED DESCRIPTION:
BACKGROUND. Parenteral nutrition associated cholestasis (PNAC) is a common complication of prolonged and exclusive parenteral nutrition (PN). PNAC in neonates and infants is multifactorial, including the underlying pathology and the effect of certain PN nutrients. In preterm infants, hepatic immaturity is itself, a predisposing factor. Infants subjected to major surgery are often unable to receive enteral nutrition for a long period of time, during which they require exclusive PN. After that, enteral nutrition is slowly introduced alongside with the reduction of the PN. In major surgery for congenital malformations of the digestive tract, additional risk factors for PNAC are the absence of enteral nutrition, intestinal bacterial translocation and sepsis. Jejunal atresia and gastroschisis are independent risk factors for PNAC. In short bowel syndrome, changes in the bile acids enterohepatic cycle may also contribute to PNAC.

Intravenous lipid emulsions (ILE) used in PN may promote PNAC or protect against it depending on their composition. Phytosterols contained in ILE have been implicated in PNAC in newborns by disrupting bile-acid homeostasis. High intakes of soy-based fatty acids (FA) n-6 from ILE, especially palmitate, may contribute to PNAC since these are precursors of arachidonic acid, a pro-inflammatory mediator.

Medium chain triglycerides (MCT) may have a hepatic protective effect. Hence, ILE containing relatively high amounts of MCT, such as Lipofundin® (B. Braun) theoretically might be advantageous in protecting against PNAC. Long chain triglycerides (LCT) of n-3 family may protect from PNAC thorough its anti-inflammatory activity. The Omegaven® (Fresenius Kabi), exclusively based on LCT n-3 has proved to prevent and reverse PNAC in neonates.

In several new-generation emulsions, including SMOFlipid® (Fresenius Kabi), the reported α-tocopherol content is up to 4- to 5-fold higher than the alpha-tocopherol content of soy-oil emulsions. The α-tocopherol isoform acts as an antioxidant, preventing lipid peroxidation attributable to the high content of long-chain polyunsaturated fatty acid (LC-PUFA).

The ILE Lipofundin® (B Braun), is composed of 50% LCT (soybean oil) and 50% MCT (coconut oil). The other new generation ILE SMOFlipid® (Fresenius Kabi) is composed of 30% LCT n-6 (soybean oil), 30% MCT (coconut oil), 25% monounsaturated fatty acids (olive oil), 15% LCT n-3 (fish oil) and α-tocopherol.

A systematic review found lower bilirubin levels in children with intestinal failure and other conditions receiving parenteral n-3 ILE compared with n-6 ILE. However, it was concluded that current data is insufficient to support the use of parenteral n-3 ILE in children, suggesting further trials examining long-term clinical outcomes and harms.

Among several studies comparing the effect of different ILEs in PNAC in children, only the retrospective study by Pischler et al. (2014) compared SMOFlipid® with Lipofundin®. This study included 127 children aged 0-16 years, including 34 premature infants and 59 children with surgical conditions, including necrotizing enterocolitis.

Until 2011 only Lipofundin® had been used for PN in the the medical-surgical neonatal intensive care unit (NICU) of the Hospital Dona Estefânia. The further availability of SMOFlipid® led the investigators to compare the effect of both ILE on the liver tests associated with PNAC of neonates subjected to corrective surgery for major congenital abnormalities, since to the best of our knowledge no prospective study has made this comparison specifically in this population.

OBJECTIVE. To compare the incidence and severity of PNAC in term and near-term infants subjected to corrective surgery for congenital abnormalities and needing prolonged PN using the ILE SMOFlipid® or Lipofundin®. The investigators hypothesise that the use of SMOFlipid® may be more protective from PNAC than Lipofundin.

METHODS. Design: single-center, randomized, controlled and double-blinded trial: prescribing physicians were unaware of the type of ILE administered and the pharmacist who prepared and randomized the individuals to the interventions was not aware of the liver status of the participants. Simple randomization was performed by the same pharmacist (MLR) using a computer generated random number table.

Were considered eligible every consecutive neonate admitted in the NICU, with gestational age of 34 weeks or over, requiring corrective surgery of congenital anomaly of the digestive tract or indirectly affecting the digestive tract (eg, diaphragmatic hernia). Recruitment occurred in the first 48 hours after birth, if PN with ILE was initiated within the first 48 hours after birth.

Main variables recorded:

* Weekly measurement of serum: total bilirubin, conjugated bilirubin, GGT, alanine -aminotransferase (ALT) and aspartate aminotransferase (AST), alkaline phosphatase and triglycerides.
* Daily parenteral lipid intake (g/Kg)
* Reasons for reducing or stopping ILE

Secondary variables recorded:

* Gestational age, birth weight, prenatal diagnosis of congenital abnormalities
* Main and secondary diagnoses
* Major surgery (date/ day of life)
* Events, especially infectious events (date/ day of life)
* Enteral feeding initiation (date/ day of life)
* Enteral feeding: type of feeding and mode of administration. The percent of enteral intake in relation to daily fluid intake was recorded (date/ day of life): 0-50% and full enteral feeding.
* Daily weight (g)
* Weekly length (cm) and head circumference (cm)
* Weekly or every 2 weeks measurement of serum: total blood count, ionogram, calcium, phosphorus and magnesium

Potential confounders affecting the liver function:

* Sepsis according to described criteria
* Phenobarbital for treatment abstinence syndrome secondary to sedative and analgesic drugs used during the postsurgical period
* Use of ursodeoxycholic acid

Parenteral nutrition protocol based on the National Consensus for Neonatal PN . Whenever possible PN with ILE is initiated within the first 24 hours after birth. As the Pharmacy Service of the Hospital is not available for preparing individualized PN during weekends, infants admitted during this period have initiated a standard solution containing only glucose, calcium and aminoacids. Thereafter, all patients receive a similar aminoacid, glucose, electrolyte and vitamins PN solution plus ILE (SMOFlipid® or Lipofundin®).

ILE is reduced to 0.5-1.5g/kg/d if:

Hypertriglyceridemia (> 250 mg / dL) Hyperglycemia (> 150 mg / dL) Unconjugated bilirubin > 12 mg/dL Acute phase of sepsis Pulmonary hypertension If cholestasis appeared, ILE is restricted to 2-2.5 g/kg/d, the amino acids restricted to 2-2.5 g/kg/d and glucose limited to 12 mg/kg/minute Enteral nutrition protocol is the same in both groups. Minimal enteral feeding is initiated when bowel sounds are audible, and significant abdominal distention and bilious or bloody gastric residuals are absent. Initially, feeds are administered continuously, and changed to bolus feeding as soon as infants can tolerate it. Mother's milk is preferred. However, depending on the patient's condition semi-elemental (Pepti-Junior®, Danone) or elemental formula (Neocate®, Nutricia) may be preferred. Later on, these formulas are replaced with mother's milk as soon as tolerated, or if mother's milk is insufficient or unavailable, preterm formula (Miltina Prem®, Humana GmbH, Germany) may be used in preterms or infant formula (Nan 1®, Nestlé) in full-term infants.

Data collection and storage: Excel® calculation table (Microsoft Office 2007®). Statistical analysis with the support of the Research Unit of Centro Hospitalar de Lisboa Central. Categorical data were presented as frequencies (percentages), and continuous variables as mean and standard deviation (SD) or median and inter-quartile range (25th percentile-75th percentile), as appropriate.

Mixed effects regression models were used to take into account the correlation structure between measures in time. Crude and adjusted odds-ratios with corresponding 95% confidence intervals were calculated.

The level of significance was α = 0.05. Data analysis was performed using the software SPSS 22.0 (SPSS for Windows, Rel. 22.0.1. 2013. SPSS Inc., Chicago, Il, EUA) and Stata (StataCorp. 2013. Stata Statistical Software: Release 13. College Station, TX: StataCorp LP.).

Measures of outcome: Cholestasis and cholestasis severity incidence rates and associated 95% confidence intervals will be accessed for each intervention group.

Cholestasis and severe cholestasis incidence rates will be compared by calculating relative risks and the Number Needed to Harm (NNH) in association with their 95% confidence intervals.

Relative efficacy measures (hazard ratios) and possibly odds ratios will be used if group homogeneity is found.

Identification of confounders using multivariate analysis in logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* neonates admitted in the NICU,
* gestational age of 34 weeks or over,
* undergoing corrective surgery of congenital anomaly of the digestive tract or indirectly affecting the digestive tract (eg, diaphragmatic hernia)
* initiation of PN with ILE within the first 48 hours after birth.

Exclusion Criteria:

* pre-natal or early neonatal (within the first 72 hours after birth) diagnoses of congenital or acquired hepato-biliary disease, such as biliary atresia, choledochal cyst, inborn errors of metabolism, intra-hepatic familial cholestasis, infectious hepatitis, neonatal idiopathic hepatitis, biliary lithiasis and abnormalities of liver function tests .
* later neonatal diagnoses of any above mentioned pathology.
* other congenital conditions affecting the liver function, such as meconium ileus associated with cystic fibrosis.
* treatment with ursodeoxycholic acid,
* interruption of PN for more than 48 hours for any reason, except for the postsurgical period after corrective surgery of the main condition,
* transference to another unit before completing 7 days of PN.

Ages: 12 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Incidence of cholestasis | From recruitment to full enteral feeding per mouth (up to 90 postnatal days)
  Conjugated serum bilirubin >1 mg/dl (34 mmol/L) (Moyer, 2004).

SECONDARY OUTCOMES:
Severity of cholestasis | From recruitment to full enteral feeding per mouth (up to 90 postnatal days)
  The severity of cholestasis was evaluated by the magnitude of the serum conjugated bilirubin and serum γ-glutamyltranspeptidase (GGT).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Pereira-da-Silva, MD, PhD, Principal Investigator — Neonatal Intensive Care Unit, Hospital Dona Estefania, Centro Hospitalar de Lisboa Central

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burrin DG, Ng K, Stoll B, Saenz De Pipaon M. Impact of new-generation lipid emulsions on cellular mechanisms of parenteral nutrition-associated liver disease. Adv Nutr. 2014 Jan 1;5(1):82-91. doi: 10.3945/an.113.004796. PMID 24425726
- [Background] Carter BA, Taylor OA, Prendergast DR, Zimmerman TL, Von Furstenberg R, Moore DD, Karpen SJ. Stigmasterol, a soy lipid-derived phytosterol, is an antagonist of the bile acid nuclear receptor FXR. Pediatr Res. 2007 Sep;62(3):301-6. doi: 10.1203/PDR.0b013e3181256492. PMID 17622954
- [Background] Christensen RD, Henry E, Wiedmeier SE, Burnett J, Lambert DK. Identifying patients, on the first day of life, at high-risk of developing parenteral nutrition-associated liver disease. J Perinatol. 2007 May;27(5):284-90. doi: 10.1038/sj.jp.7211686. Epub 2007 Mar 8. PMID 17344923
- [Background] Deckelbaum RJ. Intravenous lipid emulsions in pediatrics: time for a change? J Pediatr Gastroenterol Nutr. 2003 Aug;37(2):112-4. doi: 10.1097/00005176-200308000-00004. No abstract available. PMID 12883292
- [Background] Driscoll DF, Bistrian BR, Demmelmair H, Koletzko B. Pharmaceutical and clinical aspects of parenteral lipid emulsions in neonatology. Clin Nutr. 2008 Aug;27(4):497-503. doi: 10.1016/j.clnu.2008.05.003. Epub 2008 Jun 26. No abstract available. PMID 18582994
- [Background] Ekema G, Falchetti D, Boroni G, Tanca AR, Altana C, Righetti L, Ridella M, Gambarotti M, Berchich L. Reversal of severe parenteral nutrition-associated liver disease in an infant with short bowel syndrome using parenteral fish oil (Omega-3 fatty acids). J Pediatr Surg. 2008 Jun;43(6):1191-5. doi: 10.1016/j.jpedsurg.2008.01.005. PMID 18558205
- [Background] Furst P, Kuhn KS. Fish oil emulsions: what benefits can they bring? Clin Nutr. 2000 Feb;19(1):7-14. doi: 10.1054/clnu.1999.0072. No abstract available. PMID 10700528
- [Background] Goulet O, Ruemmele F. Causes and management of intestinal failure in children. Gastroenterology. 2006 Feb;130(2 Suppl 1):S16-28. doi: 10.1053/j.gastro.2005.12.002. PMID 16473066
- [Background] Kelly DA. Liver complications of pediatric parenteral nutrition--epidemiology. Nutrition. 1998 Jan;14(1):153-7. doi: 10.1016/s0899-9007(97)00232-3. PMID 9437702
- [Background] Schwab F, Geffers C, Barwolff S, Ruden H, Gastmeier P. Reducing neonatal nosocomial bloodstream infections through participation in a national surveillance system. J Hosp Infect. 2007 Apr;65(4):319-25. doi: 10.1016/j.jhin.2006.12.020. Epub 2007 Mar 12. PMID 17350730
- [Background] Teitelbaum DH, Tracy T. Parenteral nutrition-associated cholestasis. Semin Pediatr Surg. 2001 May;10(2):72-80. doi: 10.1053/spsu.2001.22386. PMID 11329608
- [Result] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188
- [Result] Kaufman SS. Prevention of parenteral nutrition-associated liver disease in children. Pediatr Transplant. 2002 Feb;6(1):37-42. doi: 10.1034/j.1399-3046.2002.1o061.x. PMID 11906641
- [Result] Koletzko B, Goulet O. Fish oil containing intravenous lipid emulsions in parenteral nutrition-associated cholestatic liver disease. Curr Opin Clin Nutr Metab Care. 2010 May;13(3):321-6. doi: 10.1097/MCO.0b013e3283385407. PMID 20393276
- [Result] Lee SI, Valim C, Johnston P, Le HD, Meisel J, Arsenault DA, Gura KM, Puder M. Impact of fish oil-based lipid emulsion on serum triglyceride, bilirubin, and albumin levels in children with parenteral nutrition-associated liver disease. Pediatr Res. 2009 Dec;66(6):698-703. doi: 10.1203/PDR.0b013e3181bbdf2b. PMID 19687773
- [Result] Moyer V, Freese DK, Whitington PF, Olson AD, Brewer F, Colletti RB, Heyman MB; North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. Guideline for the evaluation of cholestatic jaundice in infants: recommendations of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2004 Aug;39(2):115-28. doi: 10.1097/00005176-200408000-00001. PMID 15269615
- [Result] Pichler J, Simchowitz V, Macdonald S, Hill S. Comparison of liver function with two new/mixed intravenous lipid emulsions in children with intestinal failure. Eur J Clin Nutr. 2014 Oct;68(10):1161-7. doi: 10.1038/ejcn.2014.118. Epub 2014 Jun 25. PMID 24961544
- [Result] Seida JC, Mager DR, Hartling L, Vandermeer B, Turner JM. Parenteral omega-3 fatty acid lipid emulsions for children with intestinal failure and other conditions: a systematic review. JPEN J Parenter Enteral Nutr. 2013 Jan;37(1):44-55. doi: 10.1177/0148607112450300. Epub 2012 Jun 8. PMID 22683686
- [Result] Van Aerde JE, Duerksen DR, Gramlich L, Meddings JB, Chan G, Thomson AB, Clandinin MT. Intravenous fish oil emulsion attenuates total parenteral nutrition-induced cholestasis in newborn piglets. Pediatr Res. 1999 Feb;45(2):202-8. doi: 10.1203/00006450-199902000-00008. PMID 10022591
- [Derived] Pereira-da-Silva L, Nobrega S, Rosa ML, Alves M, Pita A, Virella D, Papoila AL, Serelha M, Cordeiro-Ferreira G, Koletzko B. Parenteral nutrition-associated cholestasis and triglyceridemia in surgical term and near-term neonates: A pilot randomized controlled trial of two mixed intravenous lipid emulsions. Clin Nutr ESPEN. 2017 Dec;22:7-12. doi: 10.1016/j.clnesp.2017.08.007. Epub 2017 Aug 26. PMID 29415837